CLINICAL TRIAL: NCT07234422
Title: A Registry-Based Randomised Controlled Trial With Heart 4 Data - SELEnium and CoQ10 NuTrition for Heart Failure: H4D-SELEQT-HF
Brief Title: The SELEQT-HF (SELEnium and CoQ10 NuTrition for Heart Failure) Study Will Evaluate the Effect of Adding Selenium/and coQ10 on Top of Standard HF Therapy in Patients With HF and Will do so Using a Pragmatic, Registry Based Randomized Controlled Trial in the Netherlands.
Acronym: SELEQT-HF
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Netherlands Heart Institute (Other)
Collaborators: University Medical Center Groningen (Other); ZonMw: The Netherlands Organisation for Health Research and Development (Other); Hartstichting (Unknown); Pharma Nord (Industry); WCN (Werkgroep Cardiologische centra Nederland) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NL87982.042.24; METc 2025/02 (Other: METc UMC Groningen)
Record Dates: First submitted 2025-11-14; First posted 2025-11-18 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Heart Failure
Keywords: heart failure; selenium; coQ10; registry based randomized clinical trial
MeSH Terms: conditions — Heart Failure | interventions — Selenium; coenzyme Q10

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Selenium/CoQ10 (Experimental): Oral dosage of twice daily Selenium/CoQ10 (2 x 100 μg selenium tablets (SelenoPrecise 100 μg, Pharma Nord, Denmark) and 2 x 100 mg Q10 capsules (Bio-Quinon 100 mg B.I.D, Pharma Nord, Denmark)
  Interventions: Dietary Supplement: Selenium/CoQ10
- Placebo (Placebo Comparator)
  Interventions: Drug: Matching Placebo (B)

INTERVENTIONS:
Dietary Supplement: Selenium/CoQ10 — Oral dosage of twice daily Selenium/CoQ10 (2 x 100 μg selenium tablets (SelenoPrecise 100 μg, Pharma Nord, Denmark) and 2 x 100 mg Q10 capsules (Bio-Quinon 100 mg B.I.D, Pharma Nord, Denmark)
  Arms: Selenium/CoQ10
Drug: Matching Placebo (B) — Matching Placebo
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to learn whether taking selenium and coenzyme Q10 (CoQ10) can reduce HF related events and deaths related to cardiovascular disease.

Researchers will compare selenium-CoQ10 supplements with a placebo to see if the supplements improve heart health and patient outcomes.

Participants will:

Receive either selenium-CoQ10 or placebo in addition to their usual heart failure treatment

Attend standard clinical visits according to routine clinical care.

The study will include 1,100 adults with chronic heart failure. Selenium and CoQ10 are natural nutrients with no known health risks. If effective, this supplement could provide a safe new way to improve outcomes for people with heart failure.

DETAILED DESCRIPTION:
This randomized controlled trial will be a pragmatic registry based clinical trial (RBRCT), using existing infrastructure on quality reporting of cardiovascular disease management in the Netherlands. This registration platform (Netherlands Heart Registration (NHR) forms the basis of incorporating information of patients with HF in hospitals in the Netherlands. Using the data gathered through this registry, these data will serve as source documentation for the electronic case report form of the current RBRCT and requires only limited additional information. Through the same system, randomization, (Serious) adverse event reporting, endpoint reporting and investigational product allocation will be conducted. Investigational product (selenium/CoQ10 supplementation or placebo) will be distributed from central pharmacy to the home of the patient. Apart from telephone calls at 6 months after randomization and every 12 months thereafter, there will be no study visits and the data gathering will be conducted through routine clinical care and registrations that are already in place. SELEQT-HF is an event driven RBRCT, with an expected median follow up of 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Outpatients with chronic HF, NYHA II - ambulatory IV
* Serum NT-proBNP concentrations >600 pg/mL (71 pmol/L) if in sinus rhythm; >1000pg/mL (118 pmol/L) if in Atrial fibrillation*

Exclusion Criteria:

* History of myocardial infarction, myocarditis, percutaneous intervention, cardiac surgery or stroke <30 days
* The presence of a mechanical assist device
* Scheduled for mechanical assist device or heart transplant
* Other non-cardiac conditions with limited life expectancy (<1 year)
* Amyloid, hypertrophic obstructive or constrictive cardiomyopathy
* End stage kidney disease for which chronic intermittent peritoneal or haemodialysis
* Unable to sign informed consent
* (Unwilling to stop) use of over the counter supplements coQ10/selenium
* Peanut and/or soy allergy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1100 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2030-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Composite of repeated HF hospitalization, repeated urgent HF visits and cardiovascular death | ongoing, up to ~30 months
  Total (first and subsequent) HF hospitalizations, urgent visits for HF visits and cardiovascular deaths with selenium/coQ10 compared to placebo.

SECONDARY OUTCOMES:
Total number of events of (repeated) HF hospitalization and (repeated) urgent HF visits | ongoing, up to ~30 months
  Total number of (repeated) HF hospitalization and (repeated) urgent HF visits
Time to death from any cause | ongoing, up to ~30 months
  time to death from any cause with selenium/coQ10 compared to placebo
Time to cardiovascular death | ongoing, up to ~30 months
  Time to cardiovascular death with selenium/coQ10 compared to placebo

OTHER OUTCOMES:
Total number of (repeated) all cause hospitalizations | ongoing, up to ~30 months
  Total number of (repeated) all cause hospitalizations with selenium/coQ10 compared to placebo
Total number of (repeated) unscheduled cardiovascular hospital visits | ongoing, up to ~30 months
  Total number of (repeated) unscheduled cardiovascular hospital visits with selenium/coQ10 compared to placebo
Total days alive out of hospital | ongoing, up to ~30 months
  Total days alive out of hospital with selenium/coQ10 compared to placebo
Side effects associated with study supplement | ongoing, up to 30 months
  Side effects associated with study supplement

CONTACTS AND LOCATIONS:
Overall Officials: Peter van der Meer, prof dr, Principal Investigator — University Medical Center Groningen; Jeroen Schaap, MD,PhD, Principal Investigator — Amphia Hospital Breda
Locations (7):
- Netherlands (7):
  - Noordwest Ziekenhuisgroep, Alkmaar
  - AUMC, Amsterdam
  - Amphia Ziekenhuis, Breda
  - Catharina ziekenhuis Eindhoven, Eindhoven
  - TREANT, Emmen
  - University Medical Center Groningen, Groningen
  - St Antonius ziekenhuis, Nieuwegein

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Alehagen U, Johansson P, Bjornstedt M, Rosen A, Dahlstrom U. Cardiovascular mortality and N-terminal-proBNP reduced after combined selenium and coenzyme Q10 supplementation: a 5-year prospective randomized double-blind placebo-controlled trial among elderly Swedish citizens. Int J Cardiol. 2013 Sep 1;167(5):1860-6. doi: 10.1016/j.ijcard.2012.04.156. Epub 2012 May 23. PMID 22626835
- [Background] Mortensen SA, Rosenfeldt F, Kumar A, Dolliner P, Filipiak KJ, Pella D, Alehagen U, Steurer G, Littarru GP; Q-SYMBIO Study Investigators. The effect of coenzyme Q10 on morbidity and mortality in chronic heart failure: results from Q-SYMBIO: a randomized double-blind trial. JACC Heart Fail. 2014 Dec;2(6):641-9. doi: 10.1016/j.jchf.2014.06.008. Epub 2014 Oct 1. PMID 25282031
- [Background] Bomer N, Grote Beverborg N, Hoes MF, Streng KW, Vermeer M, Dokter MM, IJmker J, Anker SD, Cleland JGF, Hillege HL, Lang CC, Ng LL, Samani NJ, Tromp J, van Veldhuisen DJ, Touw DJ, Voors AA, van der Meer P. Selenium and outcome in heart failure. Eur J Heart Fail. 2020 Aug;22(8):1415-1423. doi: 10.1002/ejhf.1644. Epub 2019 Dec 6. PMID 31808274
- [Background] Folkers K, Vadhanavikit S, Mortensen SA. Biochemical rationale and myocardial tissue data on the effective therapy of cardiomyopathy with coenzyme Q10. Proc Natl Acad Sci U S A. 1985 Feb;82(3):901-4. doi: 10.1073/pnas.82.3.901. PMID 3856239
- [Background] McKeag NA, McKinley MC, Harbinson MT, McGinty A, Neville CE, Woodside JV, McKeown PP. Dietary Micronutrient Intake and Micronutrient Status in Patients With Chronic Stable Heart Failure: An Observational Study. J Cardiovasc Nurs. 2017 Mar/Apr;32(2):148-155. doi: 10.1097/JCN.0000000000000322. PMID 26829748
- See also: ZonMW project page SELEQT-HF — https://projecten.zonmw.nl/nl/project/selenium-and-coq10-treatment-heart-failure-seleqt-hf-registry-based-randomised-clinical